CLINICAL TRIAL: NCT07205679
Title: Cardiovascular Performance and Exercise Response in Patients With Persistent or Permanent Atrial Fibrillation and Heart Failure Pre and Post Cardioversion or Pace and Ablate
Acronym: CPEX-CPA
Status: Not yet recruiting | Type: Observational
Sponsor: Habib Khan (Other)
Responsible Party: Sponsor-Investigator, Habib Khan, MBBS, PhD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: 125097; 125097 (Other: Health Sciences Research Ethics Board - Western University)
Record Dates: First submitted 2025-07-28; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF); Heart Failure - NYHA II - IV; Pacemaker; Cardioversion; Ablation Therapy
Keywords: Cardiopulmonary Exercise Testing
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardioversion: Patients with persistent AF and HF scheduled for cardioversion.
- Pace and Ablate: Patients with chronic AF and HF who are scheduled for P&A procedure.

SUMMARY:
Heart Failure (HF) and Atrial Fibrillation (AF) are two conditions that commonly occur together. Clinical guidelines consider a resting heart rate of 100-110 beats per minute (bpm) acceptable for patients with HF and AF while 72 bpm is considered the average in healthy populations. A higher resting heart rate indicates that the heart is working harder to meet bodily demands, and though it may be considered safe for patients with HF and AF to have a heart rate of 110 bpm, the investigators believe it is having a significant negative impact on patient quality of life and their ability to exercise. The current study will test exercise ability using a treadmill test before and after either a cardioversion, where the patient's heartbeat is reset using electric shocks, or a pace and ablate method, where the patient receives a pacemaker to regulate their heart rhythm and an ablation (intentional damaging) of the node that coordinates the beats within the heart. This will allow investigators to compare how the heart responds to exercise when the patient is on rate-control and anticoagulation medication therapy (before cardioversion or pace and ablate) and after the procedures. During exercise, the investigators will do a blood test that lets investigators know how efficiently the heart is working and record any symptoms experienced. The investigators will also collect information about the patient's quality of life. Using this information, the investigators hope to better understand whether the current standard of a resting heart rate of 100-110 bpm is ideal for patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Persistent or Permanent Atrial Fibrillation
3. HF - NYHA class II-IVA despite guideline-direct medical therapy
4. Rate controlled
5. Able to perform stress test
6. Scheduled for clinical P&A OR cardioversion

Exclusion Criteria:

1. Creatinine >180 μmol/L or eGFR <30 mL/min/1.73 m2
2. Significant valvular heart disease: Moderate to severe tricuspid regurgitation, mitral regurgitation, mitral stenosis, aortic regurgitation, aortic stenosis
3. Patients who have had a TAVI, valvular surgery, or CABG within 3 months of enrolment
4. Right ventricular systolic pressure >50mmHg
5. Existing pacemaker
6. In sinus rhythm
7. Predictable vasovagal syncope to pain and sight of blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been clinically scheduled for either a P&A or a cardioversion procedure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Exercise duration | 1 month
Peak oxygen update | 1 month
  Peak oxygen uptake achieved during a symptom-limited incremental exercise test to task failure.
B-type Natriuretic Peptide (BNP) Test | 1 month

SECONDARY OUTCOMES:
Change in maximal HR during exercise | 1 month
EuroQol (EQ-5D-5L) | 1 month
  Participants indicate abilities with respect to five dimensions of health. Higher scores indicate greater impairment.
Rate of Perceived exertion change during exercise | 1 month
V̇O2peak change | 1 month
Change in lactate threshold | 1 month
Kansas City Cardiomyopathy Questionnaire | 1 month
  Change in Kansas HF score from baseline. KCCQ is a 23-item self-administered questionnaire that measures the participant's perception of their health status, including their HF symptoms, impact on physical and social function and how their HF impacts the quality of life (QoL). KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), QoL (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status.